CLINICAL TRIAL: NCT04235998
Title: Value of Additional Upfront Systematic Lung Ultrasound in the Workup of Patients With Unilateral Pleural Effusion: A Prospective Cohort Study
Brief Title: Value of Additional Upfront Systematic Lung Ultrasound in the Workup of Patients With Unilateral Pleural Effusion
Status: Completed | Type: Observational
Sponsor: Naestved Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-789
Record Dates: First submitted 2019-12-19; First posted 2020-01-22 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Pleural Effusion; Malignant Pleural Effusion; Ultrasound
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Systematic lung ultrasound: Patients with unilateral pleural effusion of unknown course
  Interventions: Diagnostic Test: Systematic lung ultrasound

INTERVENTIONS:
Diagnostic Test: Systematic lung ultrasound — Patients will undergo a systematic lung ultrasound including review of:
  * Sonographic characteristic of effusion
  * Parietal, diaphragmatic and visceral pleura
  * Pleural nodules
  * Lung parenchyma
  * Extra pulmonary findings: Hepatic pathology, enlarged lymph nodes of the neck and a cardiac assessment.

SUMMARY:
The value of lung ultrasound in the work up of pleural effusion (fluid in between the thin doublet layered film surrounding the lungs) is unknown. The researchers will perform a systematic lung ultrasound scan including a scan for extra thoracic metastasis (spread of cancer to other organs) in the lymphnodes of the neck and metastasis lever in 56 patients one-sided pleural effusion. The researchers will measure if the interventions change the diagnostic plan for the patient and leads to faster diagnostics of the underlying course.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Unilateral pleural effusion of unknown course.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Bilateral pleural effusions.
* Known cause of pleural effusions.
* Life expectancy <3 months.
* Inability to understand written or spoken Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Pleura Clinic (an outpatient clinic in the Department of Pulmonary Disease, Næstved Sygehus, on of two regional centers for work up of pulmonary malignancy ) from the general practitioner or from other hospital departments both Næstved Sygehus and other hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Proportion of cases where systematic lung ultrasound (LUS) change the planned diagnostic process for patients with unilateral pleural effusion. | 26 weeks post procedure
  Information found in electronic patient files. Comparison of diagnostics planned before systematic ultrasound and diagnostics planned after systematic ultrasound. Measured in proportion of included patients

SECONDARY OUTCOMES:
Characteristics of ultrasonic findings with additional systematic LUS. | Day 1, within 30 minutes after the end of procedure
  Characteristics is recorded in the ultrasound protocol
Proportion of cases where findings of clinical importance on systematic LUS were not identified at the initial contrast-enhanced CT thorax or PET-CT | Day 1 within 30 minutes after the end of procedure
  CT thorax and PET-CT (as assessed by radiologist or clinician at the initial planning of diagnostic work-up)
Proportion of cases where the change in the diagnostic process after LUS provide a diagnose | 26 weeks post procedure
  Information found in electronic patient files.
The patient experienced pain during procedure score | Day 1 within 30 minutes after the end of procedure
  Measured by a VAS (Visual Analogue Scale) scale 0-10, 0 being no pain, 10 being the worse pain
Patient experienced time consumption | Day 1 within 30 minutes after the end of procedure
  Measured by a 3-point Likert scale , scale1-3, 1 being not time consuming at all, 3 being very time consuming
The patients willingness to have the same examination again in the future if necessary | Day 1within 30 minutes after the end of procedure
  Measured by a 5-point Likert scale, scale 1-5, 1 being definitely willing to have the examination again, 5 being definitely not willing to have the examination again
Mean extra time spend on systematic LUS compared to conventional US for guidance of thoracentesis | Day 1 within 30 minutes after the end of procedure
  Measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Bødtger, MD, PhD, Principal Investigator — Department of Pulmonary Medicin, Næstved Sygehus
Locations (1):
- Næstved Sygehus, department of pulmonary medicine, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No